CLINICAL TRIAL: NCT05779904
Title: DNA Methylation, Microbiome Profile, Nutritional Status, and Developmental Outcomes of Stunted and Non-stunted Children Growing up During Covid-19 Pandemic: a Case-control Study
Brief Title: Methylation, mIcrobiome, NUtritional sTatus, and dEvelopment of Stunted Children
Acronym: MINUTES
Status: Active, not recruiting | Type: Observational
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Aberdeen (Other)
Responsible Party: Principal Investigator, Dr.Umi Fahmida, Principal Investigator, SEAMEO Regional Centre for Food and Nutrition
Other Study IDs: AASH Early Year Study
Record Dates: First submitted 2023-02-06; First posted 2023-03-22 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Stunting; Development, Child; DNA Methylation; Epigenetics; Nutrition
Keywords: Epigenetics signature; Case-control; Under-two-year-old children
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stunted (Case): In the case group, stunted children (<-2SD) (n=150) will be recruited.
- Non-stunted (Control): In the control group, non-stunted children (>-1SD) (n=150) will be recruited.

SUMMARY:
The investigators will conduct a case-control study among under-two children in Lombok Timur, West Nusa Tenggara, Indonesia. The power required to detect changes in epigenetic markers may not be sufficient in the cohort study. Therefore, specific case-control design of stunted vs non-stunted children will provide the required power to detect potential epigenetic markers which will be further investigated through targeted sequencing of the cohort study. A total of 150 stunted children will be recruited and then it will be matched with 150 non-stunted children with the same sex. The assessments for these study subjects will include: 1) The genetic and epigenetic profile of the children, gut microbiota and nutritional status (Physical component), 2) Food security, Water, Sanitation and Hygiene (WASH) and Infant and Young Child Feeding (IYCF) practices (Home-Food component), 3) Children's psychosocial care and cognitive outcome (Cognition component).

DETAILED DESCRIPTION:
This study is part of Action Against Stunting Hub, an observational cohort study aimed to build evidence based on exploring the drivers of stunting from different perspectives and understand the impact of different interventions across three countries: India, Indonesia and Senegal. This study is intended to give the overview of stunting and its determinants among under-two children growing up during period of Covid-19 pandemic in Lombok Timur, Nusa Tenggara Barat, Indonesia. Because, the power required to detect changes in epigenetic markers may not be sufficient in the cohort study, this specific case-control design of stunted vs non-stunted children will also provide the required power to detect potential epigenetic markers which will be further investigated through targeted sequencing of the cohort study. The results of this initial study are projected to support further study, especially the observational cohort study, in determining the best suited indicators to prove the interaction and/or causal mechanisms of stunting.

ELIGIBILITY:
Inclusion Criteria:

* aged 18.0 - 23.9 months
* without serious illnesses
* the mother delivered the children between 18-40 years of age
* has Sasak ethnicity, (5) recumbent length <-2SD (for stunted group) and >-1SD (for non- stunted group) from the WHO Child Growth Standards median for their age and sex at the recruitment.

Exclusion Criteria:

* twin birth
* congenital malformation
* consanguinity

Ages: 18 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 150 stunted children (case) will be recruited and then it will be matched with 150 non-stunted children (control) with the same sex. Before the screening time, data of children aged 18.0-23.9 months from Posyandu will be listed. The field team will coordinate with midwives to inform the children and their guardian to get screened. Screening for eligibility criteria will be done for all children aged 18.0-23.9 months that has listed in the previous visit. Length measurement for the children and checklist of eligibility criteria will be done during the screening time by trained enumerators. After fulfilling the eligibility criteria, the enumerators have to determine to matched children based on their gender.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Epigenetics signature related to stunting | at enrollment
  Analysis of epigenetic states (DNA methylation) will be carried out using the Illumina Infinium Methylation EPIC V.2.0 BeadChip, augmented by sequencing methodologies to provide both genome wide coverage and high-definition analysis. Epigenetic state controls gene expression and overall genome regulation at scale and the study will focus on candidate epigenetic states implicated in stunting and its corollaries alongside epigenome wide association.

SECONDARY OUTCOMES:
Child congnition outcomes (by psychologists) | at enrollment
  Cognitive development will be assessed using the full Bayley Scales of Infant and Toddler Development (BSID-4) by trained psychologists. BSID-4 consists of: Cognitive Scale (COG); Language Scale (LANG), and Motoric Scale (MOT).
  The range of Standard Score (SS) of each scale is 40-160 in which higher score means better.
Child cognition outcomes (care giver reported) | at enrollment
  Cognitive development will be assessed using the care giver reported tool, i.e., INTERGROWTH-21st Neurodevelopment assessment INTER-NDA by trained enumerators. INTER-NDA consists of: Cognitive; Fine motor; Gross motor; Language; Positive behavior; Negative behavior.
  The range of score on each scale is 0 - 100 in which higher score means better.
Gut microbiome | at enrollment
  Faecal microbiome would be analyzed using 16S RNA sequencing of the V4 region on the Illumina MiSeq platform

CONTACTS AND LOCATIONS:
Overall Officials: Umi Fahmida, Dr., Principal Investigator — SEAMEO RECFON
Locations (1):
- Seameo Recfon, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguilar-Farias N, Toledo-Vargas M, Miranda-Marquez S, Cortinez-O'Ryan A, Cristi-Montero C, Rodriguez-Rodriguez F, Martino-Fuentealba P, Okely AD, Del Pozo Cruz B. Sociodemographic Predictors of Changes in Physical Activity, Screen Time, and Sleep among Toddlers and Preschoolers in Chile during the COVID-19 Pandemic. Int J Environ Res Public Health. 2020 Dec 29;18(1):176. doi: 10.3390/ijerph18010176. PMID 33383721
- [Background] Ansari I, Raddatz G, Gutekunst J, Ridnik M, Cohen D, Abu-Remaileh M, Tuganbaev T, Shapiro H, Pikarsky E, Elinav E, Lyko F, Bergman Y. The microbiota programs DNA methylation to control intestinal homeostasis and inflammation. Nat Microbiol. 2020 Apr;5(4):610-619. doi: 10.1038/s41564-019-0659-3. Epub 2020 Feb 3. PMID 32015497
- [Background] Bosso M, Thanaraj TA, Abu-Farha M, Alanbaei M, Abubaker J, Al-Mulla F. The Two Faces of ACE2: The Role of ACE2 Receptor and Its Polymorphisms in Hypertension and COVID-19. Mol Ther Methods Clin Dev. 2020 Jun 25;18:321-327. doi: 10.1016/j.omtm.2020.06.017. eCollection 2020 Sep 11. PMID 32665962
- [Background] Burchill E, Lymberopoulos E, Menozzi E, Budhdeo S, McIlroy JR, Macnaughtan J, Sharma N. The Unique Impact of COVID-19 on Human Gut Microbiome Research. Front Med (Lausanne). 2021 Mar 16;8:652464. doi: 10.3389/fmed.2021.652464. eCollection 2021. PMID 33796545
- [Background] Campagna MP, Xavier A, Lechner-Scott J, Maltby V, Scott RJ, Butzkueven H, Jokubaitis VG, Lea RA. Epigenome-wide association studies: current knowledge, strategies and recommendations. Clin Epigenetics. 2021 Dec 4;13(1):214. doi: 10.1186/s13148-021-01200-8. PMID 34863305
- [Background] Carroll N, Sadowski A, Laila A, Hruska V, Nixon M, Ma DWL, Haines J, On Behalf Of The Guelph Family Health Study. The Impact of COVID-19 on Health Behavior, Stress, Financial and Food Security among Middle to High Income Canadian Families with Young Children. Nutrients. 2020 Aug 7;12(8):2352. doi: 10.3390/nu12082352. PMID 32784530
- [Background] Cryan JF, Dinan TG. Mind-altering microorganisms: the impact of the gut microbiota on brain and behaviour. Nat Rev Neurosci. 2012 Oct;13(10):701-12. doi: 10.1038/nrn3346. Epub 2012 Sep 12. PMID 22968153
- [Background] Development Initiatives (2018). 2018 Global Nutrition Report: Shining a light to spur action on nutrition. Bristol, UK: Development Initiatives.
- [Background] Development Initiatives Poverty Research. 2020. 2020 Global Nutrition Report: Action on equity to end malnutrition. Bristol, UK: Development Initiatives.
- [Background] Haggarty P, Hoad G, Campbell DM, Horgan GW, Piyathilake C, McNeill G. Folate in pregnancy and imprinted gene and repeat element methylation in the offspring. Am J Clin Nutr. 2013 Jan;97(1):94-9. doi: 10.3945/ajcn.112.042572. Epub 2012 Nov 14. PMID 23151531
- [Background] Haggarty, P., K. Harrison and Haggarty (2017). Population Epigenetics, Springer.
- [Background] Hannon E, Schendel D, Ladd-Acosta C, Grove J, Hansen CS, Hougaard DM, Bresnahan M, Mors O, Hollegaard MV, Baekvad-Hansen M, Hornig M, Mortensen PB, Borglum AD, Werge T, Pedersen MG, Nordentoft M; iPSYCH-Broad ASD Group; Buxbaum JD, Daniele Fallin M, Bybjerg-Grauholm J, Reichenberg A, Mill J. Variable DNA methylation in neonates mediates the association between prenatal smoking and birth weight. Philos Trans R Soc Lond B Biol Sci. 2019 Apr 15;374(1770):20180120. doi: 10.1098/rstb.2018.0120. PMID 30966880
- [Background] Harpham T, Reichenheim M, Oser R, Thomas E, Hamid N, Jaswal S, Ludermir A, Aidoo M. Measuring mental health in a cost-effective manner. Health Policy Plan. 2003 Sep;18(3):344-9. doi: 10.1093/heapol/czg041. PMID 12917276
- [Background] He J, Lu YP, Li J, Li TY, Chen X, Liang XJ, Chen WJ, Pi SN, Hocher B, Chen YP. Fetal But Not Maternal Angiotensin Converting Enzyme (ACE)-2 Gene Rs2074192 Polymorphism is Associated with Increased Risk of Being a Small For Gestational Age (SGA) Newborn. Kidney Blood Press Res. 2018;43(5):1596-1606. doi: 10.1159/000494449. Epub 2018 Oct 22. PMID 30347406
- [Background] Hoddinott J, Behrman JR, Maluccio JA, Melgar P, Quisumbing AR, Ramirez-Zea M, Stein AD, Yount KM, Martorell R. Adult consequences of growth failure in early childhood. Am J Clin Nutr. 2013 Nov;98(5):1170-8. doi: 10.3945/ajcn.113.064584. Epub 2013 Sep 4. PMID 24004889
- [Background] Huang M, Liu J, Liu K, Chen J, Wei Z, Feng Z, Wu Y, Fong M, Tian R, Wang B, Budjan C, Zhuang P, Wan G, Kong XJ. Microbiome-Specific Statistical Modeling Identifies Interplay Between Gastrointestinal Microbiome and Neurobehavioral Outcomes in Patients With Autism: A Case Control Study. Front Psychiatry. 2021 Oct 20;12:682454. doi: 10.3389/fpsyt.2021.682454. eCollection 2021. PMID 34744810
- [Background] James P, Sajjadi S, Tomar AS, Saffari A, Fall CHD, Prentice AM, Shrestha S, Issarapu P, Yadav DK, Kaur L, Lillycrop K, Silver M, Chandak GR; EMPHASIS study group. Candidate genes linking maternal nutrient exposure to offspring health via DNA methylation: a review of existing evidence in humans with specific focus on one-carbon metabolism. Int J Epidemiol. 2018 Dec 1;47(6):1910-1937. doi: 10.1093/ije/dyy153. PMID 30137462
- [Background] Littlejohn P, Finlay BB. When a pandemic and an epidemic collide: COVID-19, gut microbiota, and the double burden of malnutrition. BMC Med. 2021 Jan 28;19(1):31. doi: 10.1186/s12916-021-01910-z. PMID 33504332
- [Background] Lima RS, Rocha LPC, Moreira PR. Genetic and epigenetic control of ACE2 expression and its possible role in COVID-19. Cell Biochem Funct. 2021 Aug;39(6):713-726. doi: 10.1002/cbf.3648. Epub 2021 Jun 1. PMID 34075603
- [Background] Lozupone CA, Stombaugh J, Gonzalez A, Ackermann G, Wendel D, Vazquez-Baeza Y, Jansson JK, Gordon JI, Knight R. Meta-analyses of studies of the human microbiota. Genome Res. 2013 Oct;23(10):1704-14. doi: 10.1101/gr.151803.112. Epub 2013 Jul 16. PMID 23861384
- [Background] MAL-ED Network Investigators. Childhood stunting in relation to the pre- and postnatal environment during the first 2 years of life: The MAL-ED longitudinal birth cohort study. PLoS Med. 2017 Oct 25;14(10):e1002408. doi: 10.1371/journal.pmed.1002408. eCollection 2017 Oct. PMID 29069076
- [Background] Mansell G, Gorrie-Stone TJ, Bao Y, Kumari M, Schalkwyk LS, Mill J, Hannon E. Guidance for DNA methylation studies: statistical insights from the Illumina EPIC array. BMC Genomics. 2019 May 14;20(1):366. doi: 10.1186/s12864-019-5761-7. PMID 31088362
- [Background] Masser DR, Stanford DR, Freeman WM. Targeted DNA methylation analysis by next-generation sequencing. J Vis Exp. 2015 Feb 24;(96):52488. doi: 10.3791/52488. PMID 25741966
- [Background] McArthur, BA., Browne, D., Tough, S., and Madigan, S. (2020). Trajectories of screen use during early childhood: Predictors and associated behavior and learning outcomes. Computers in Human Behavior 113: 106501.
- [Background] Miguel PM, Pereira LO, Silveira PP, Meaney MJ. Early environmental influences on the development of children's brain structure and function. Dev Med Child Neurol. 2019 Oct;61(10):1127-1133. doi: 10.1111/dmcn.14182. Epub 2019 Feb 11. PMID 30740660
- [Background] Ministry of Health RI. 2021. Indonesia Nutritional Status Study 2021. (disseminated study through national event)
- [Background] Neumann, C., D. M. Harris and L. M. Rogers (2002). Contribution of animal source foods in improving diet quality and function in children in the developing world. Nutrition research 22(1-2): 193-220.
- [Background] Ngure FM, Reid BM, Humphrey JH, Mbuya MN, Pelto G, Stoltzfus RJ. Water, sanitation, and hygiene (WASH), environmental enteropathy, nutrition, and early child development: making the links. Ann N Y Acad Sci. 2014 Jan;1308:118-128. doi: 10.1111/nyas.12330. PMID 24571214
- [Background] Noor N, Cardenas A, Rifas-Shiman SL, Pan H, Dreyfuss JM, Oken E, Hivert MF, James-Todd T, Patti ME, Isganaitis E. Association of Periconception Paternal Body Mass Index With Persistent Changes in DNA Methylation of Offspring in Childhood. JAMA Netw Open. 2019 Dec 2;2(12):e1916777. doi: 10.1001/jamanetworkopen.2019.16777. PMID 31880793
- [Background] Nwosu BU, Lee MM. Evaluation of short and tall stature in children. Am Fam Physician. 2008 Sep 1;78(5):597-604. PMID 18788236
- [Background] Olofin I, McDonald CM, Ezzati M, Flaxman S, Black RE, Fawzi WW, Caulfield LE, Danaei G; Nutrition Impact Model Study (anthropometry cohort pooling). Associations of suboptimal growth with all-cause and cause-specific mortality in children under five years: a pooled analysis of ten prospective studies. PLoS One. 2013 May 29;8(5):e64636. doi: 10.1371/journal.pone.0064636. Print 2013. PMID 23734210
- [Background] Osendarp S, Akuoku JK, Black RE, Headey D, Ruel M, Scott N, Shekar M, Walker N, Flory A, Haddad L, Laborde D, Stegmuller A, Thomas M, Heidkamp R. The COVID-19 crisis will exacerbate maternal and child undernutrition and child mortality in low- and middle-income countries. Nat Food. 2021 Jul;2(7):476-484. doi: 10.1038/s43016-021-00319-4. Epub 2021 Jul 19. PMID 37117686
- [Background] Ozaltin E, Hill K, Subramanian SV. Association of maternal stature with offspring mortality, underweight, and stunting in low- to middle-income countries. JAMA. 2010 Apr 21;303(15):1507-16. doi: 10.1001/jama.2010.450. PMID 20407060
- [Background] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603
- [Background] Rinninella E, Raoul P, Cintoni M, Franceschi F, Miggiano GAD, Gasbarrini A, Mele MC. What is the Healthy Gut Microbiota Composition? A Changing Ecosystem across Age, Environment, Diet, and Diseases. Microorganisms. 2019 Jan 10;7(1):14. doi: 10.3390/microorganisms7010014. PMID 30634578
- [Background] Riskesdas (2018). Departemen Kesehatan Republik Indonesia, Laporan Hasil Riset Kesehatan Dasar Indonesia (Riskesdas) 2018. Jakarta, Republic of Indonesia.
- [Background] Robertson RC, Manges AR, Finlay BB, Prendergast AJ. The Human Microbiome and Child Growth - First 1000 Days and Beyond. Trends Microbiol. 2019 Feb;27(2):131-147. doi: 10.1016/j.tim.2018.09.008. Epub 2018 Oct 24. PMID 30529020
- [Background] Stephenson LS, Latham MC, Ottesen EA. Malnutrition and parasitic helminth infections. Parasitology. 2000;121 Suppl:S23-38. doi: 10.1017/s0031182000006491. PMID 11386688
- [Background] Stewart CP, Iannotti L, Dewey KG, Michaelsen KF, Onyango AW. Contextualising complementary feeding in a broader framework for stunting prevention. Matern Child Nutr. 2013 Sep;9 Suppl 2(Suppl 2):27-45. doi: 10.1111/mcn.12088. PMID 24074316
- [Background] Sudfeld CR, McCoy DC, Danaei G, Fink G, Ezzati M, Andrews KG, Fawzi WW. Linear growth and child development in low- and middle-income countries: a meta-analysis. Pediatrics. 2015 May;135(5):e1266-75. doi: 10.1542/peds.2014-3111. Epub 2015 Apr 6. PMID 25847806
- [Background] Tian Y, Morris TJ, Webster AP, Yang Z, Beck S, Feber A, Teschendorff AE. ChAMP: updated methylation analysis pipeline for Illumina BeadChips. Bioinformatics. 2017 Dec 15;33(24):3982-3984. doi: 10.1093/bioinformatics/btx513. PMID 28961746
- [Background] UNICEF. COVID-19 and Children in Indonesia.An Agenda for Action to Address Socio-Economic Challenges. 11 May 2020
- [Background] Walker SP, Chang SM, Powell CA, Simonoff E, Grantham-McGregor SM. Early childhood stunting is associated with poor psychological functioning in late adolescence and effects are reduced by psychosocial stimulation. J Nutr. 2007 Nov;137(11):2464-9. doi: 10.1093/jn/137.11.2464. PMID 17951486
- [Background] Williams AM, Suchdev PS. Assessing and Improving Childhood Nutrition and Growth Globally. Pediatr Clin North Am. 2017 Aug;64(4):755-768. doi: 10.1016/j.pcl.2017.03.001. PMID 28734508
- [Background] Ye J, Wu W, Li Y, Li L. Influences of the Gut Microbiota on DNA Methylation and Histone Modification. Dig Dis Sci. 2017 May;62(5):1155-1164. doi: 10.1007/s10620-017-4538-6. Epub 2017 Mar 24. PMID 28341870
- [Background] Yu G, Wang LG, Han Y, He QY. clusterProfiler: an R package for comparing biological themes among gene clusters. OMICS. 2012 May;16(5):284-7. doi: 10.1089/omi.2011.0118. Epub 2012 Mar 28. PMID 22455463
- [Background] Zemrani B, Gehri M, Masserey E, Knob C, Pellaton R. A hidden side of the COVID-19 pandemic in children: the double burden of undernutrition and overnutrition. Int J Equity Health. 2021 Jan 22;20(1):44. doi: 10.1186/s12939-021-01390-w. PMID 33482829